CLINICAL TRIAL: NCT05457842
Title: A Phase 2 Open-label, Dose-finding Study to Determine the Optimal Dose for Lymph Node Visualization Using ASP5354 in Participants With Breast Cancer or Melanoma Undergoing Sentinel Lymph Node Biopsy
Brief Title: A Study to Find the Best Dose of ASP5354 to Show Lymph Nodes in People With Breast Cancer or Melanoma During Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company's strategic decision
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 5354-CL-1201
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sentinel Lymph Node Biopsy; Breast Cancer; Melanoma
Keywords: ASP5354; pudexacianinium chloride; SLN; Breast Cancer; Melanoma
MeSH Terms: conditions — Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASP5354 0.2 mg (Experimental): Participant received a single dose of 0.2 milligrams (mg) intradermal injection of ASP5354 on day 1.
  Interventions: Drug: pudexacianinium chloride

INTERVENTIONS:
Drug: pudexacianinium chloride — Intradermal injection
  Other Names: ASP5354

SUMMARY:
This study was for women with breast cancer and for adults with melanoma. Breast cancer was a type of cancer when cells in the breast turn into cancer cells, which might grow out of control. Melanoma was a type of skin cancer that starts in cells called melanocytes. These cells made a substance called melanin which gives the skin its color. In this study, people had surgery to remove the lymph node closest to the site of their cancer. This lymph node was called the sentinel node. This was done to check if the cancer had spread from the original site to the sentinel node. This procedure was called a sentinel node biopsy.

This study provided more information on a potential new dye, called ASP5354, used in sentinel node biopsies. ASP5354 helped to show the lymph nodes more clearly during surgery. This helped the surgeon find the lymph node closest to the site of the cancer (sentinel node).

The main aim of the study was to find the best dose of ASP5354 that clearly showed the lymph nodes during surgery. This was an open-label study. That means each person in the study and the study doctors knew that person received ASP5354.

Each person only received 1 dose of ASP5354.

People that wanted to take part in the study were checked by a study doctor. This was on a separate visit before their surgery. Before surgery, people who took part in the study were asked if they had any other medical problems. They had a physical exam, an ECG to check their heart rhythm, and had their vital signs checked (blood pressure, pulse rate, and breathing rate). Other checks included some blood and urine samples taken for laboratory tests.

During surgery, a study surgeon injected ASP5354 near the cancer site. They recorded how clearly they could see the lymph nodes. Some blood samples were taken for laboratory tests and an ECG was done. After their surgery, people were asked if they have any other medical problems.

People returned to the hospital 9 days later for a check-up. The check-up included a physical exam, an ECG to check their heart rhythm, and a check of their vital signs (blood pressure, pulse rate, and breathing rate). Other checks included some blood samples taken for laboratory tests. People were asked if they had any medical problems and asked to complete a feedback survey.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been diagnosed with localized breast cancer (female only, stage 1 to 2, N0 and M0) or melanoma (stage 1 to 2, N0 and M0) and is scheduled to undergo surgical intervention for systemic lymph node (SLN) detection and removal using Technetium-99m sulfur colloid or Lymphoseek as part of Standard of Care (SOC).
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final study treatment administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final study treatment administration.
* Female participant must not donate ova starting at first dose of Investigational Product (IP) and throughout the study period and for 30 days after final study treatment administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use of contraception throughout the treatment period and for 30 days after final study treatment administration.
* Male participant must not donate sperm during the treatment period and for 30 days after final study treatment administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final study treatment administration.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has had prior lymph node (LN) surgery in the area where LN detection is needed.
* Participant has had prior LN radiation in the area where LN detection is needed.
* Participant has had prior neo-adjuvant chemotherapy.
* Participant has definitive LN metastases.
* Participant has metastatic cancer.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP5354, indocyanine green (ICG) or any components of the formulation used.
* Participant has had previous exposure to ASP5354.
* Participant has moderate to severe cardiac disease that limits daily functioning (New York Heart Association Class III-IV) or other medical conditions that would impact safety or study compliance.
* Participant has a resting heart rate <= 45 beats per minute (bpm) or >=115 bpm, systolic blood pressure >=160 mm Hg or diastolic blood pressure >= 100 mm Hg within 1 week prior to IP administration. If the blood pressure exceeds the limits above, repeat readings can be taken. Participant who has adequately controlled blood pressure is eligible.
* Participant has any of the screening laboratory values outside of the protocol specification criteria.
* Participant has received ICG, other near-infrared fluorescence (NIR-F) imaging agents, Blue dye (e.g., methylene blue or isosulfan blue) or magtrace within 2 weeks prior to IP administration.
* Participant has active alcohol abuse or illicit drug use (non-prescription or over-the-counter medications). Participant should not have consumed any alcohol or illicit drug (excluding cannabidiol products) within 24 hours of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only for breast cancer segment
Enrollment: 1 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Inc
Locations (1):
- UCI Irvine Health-Chao Family Comprehensive Cancer Center Cancer, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant with breast cancer or melanoma scheduled to undergo sentinel lymph node (SLN) biopsy.
Pre-assignment Details: Female participants ≥ 18 years of age diagnosed with localized breast cancer (stage 0 to 2,N0 and M0) or melanoma (stage 1 to 2, N0 and M0) scheduled to undergo surgical intervention for SLN detection and removal using technetium-99m sulfur colloid (Tc-99mSC) or Lymphoseek as part of standard of care (SOC).
Groups:
- ASP5354 0.2 Milligrams (mg): Participant received a single dose of 0.2 mg intradermal injection of ASP5354 on day 1.
Period: Overall Study
Arm/Group | ASP5354 0.2 Milligrams (mg)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): Participant enrolled and received study Investigational product (IP).
Groups:
- ASP5354 0.2 mg: Participant received a single dose of 0.2 mg intradermal injection of ASP5354 on day 1.
Arm/Group | ASP5354 0.2 mg
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Optimal Dose of ASP5354 for Lymph Node (LN) Visualization
Description: The optimal dose was defined as the dose that provided a better visualization compared with lower doses and a comparable visualization to the next higher dose. In the case where 2 doses performed equally, the lower dose was selected. Cumulative visualization data of the LNs from all treated participants was used for optimal dose determination. The optimal dose was determined by the Visualization Review Committee (VRC) using data from the following assessments: LN tissue visualized (Y/N), visualized tissue is lymphatic in origin based on pathologic confirmation, Likert Scale determination of the intensity of fluorescence, and proportion of identified LN with histopathologic confirmation of LN tissue by ASP5354 compared with standard of care (SOC) treatment.
Time Frame: Day 1
Population: FAS
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | ASP5354 0.2 mg
Number analyzed (Participants) | 1
milligrams (mg) | NA — With 1 participant enrolled, the optimal dose could not be recorded.

2. Secondary Outcome: Percentage of Participants With at Least 1 LN Detected Using ASP5354
Description: The visualization of at least 1 LN with histopathologic confirmation is assessed by using a binary "Yes" or "No" question. Those participants with "Yes" as response was reported.
Time Frame: Day 1 up to day 10
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | ASP5354 0.2 mg
Number analyzed (Participants) | 1
percentage of participants | 100

3. Secondary Outcome: Percentage of Identified LN Tissue by ASP5354 Compared With SOC Treatment
Description: The percentage of identified LN with ASP5354 will be compared with SOC treatment with either Tc-99mSC or Lymphoseek, through histopathologic confirmation.
Time Frame: Day 1 up to day 10
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of lymph nodes
Units Other Than Participants: lymph nodes
Arm/Group | ASP5354 0.2 mg
Number analyzed (Participants) | 1
Number analyzed (lymph nodes) | 3
percentage of lymph nodes | 100.0 [NA to NA] — Due to low number of events , upper and lower level of 95% CI were not reported.

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An AE was considered "serious" if, it resulted in any of the following outcomes: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly, or birth defect; requires inpatient hospitalization; or leads to prolongation of hospitalization; other medically important events. TEAE was defined as an AE observed after starting administration of the study drug.
Time Frame: From first dose up to day 10
Population: Safety Analysis Set (SAF): Participant enrolled and received study IP.
Measure: Number; unit: Participants
Arm/Group | ASP5354 0.2 mg
Number analyzed (Participants) | 1
Participants
  TEAE | 0
  SAE | 0

5. Secondary Outcome: Plasma Concentration of ASP5354
Description: Plasma concentration of ASP5354. The Lower limit of quantification (LLOQ) was defined as 1.00 nanograms per milliliter (ng/mL). Measured values below the LLOQ were expressed as <LLOQ and not reported.
Time Frame: Predose, approximately 10 minutes, 30 minutes, 60 minutes postdose, and at the end of surgery (day 1)
Population: Pharmacokinetic analysis set: All participants who received at least 1 dose of IP for which at least 1 plasma concentration data were available with the time of dosing and sampling.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ASP5354 0.2 mg
Number analyzed (Participants) | 1
ng/mL
  Predose | NA (NA) — Data was not reported as it was <LLOQ.
  10 minutes post dose | 1.13
  30 minutes post dose | 1.75
  60 minutes post dose | 1.66
  End of surgery post dose | 1.21

ADVERSE EVENTS:
Time Frame: From first dose up to 10 days
Description: SAF
Arm/Group | ASP5354 0.2 mg
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT05457842/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT05457842/SAP_001.pdf